CLINICAL TRIAL: NCT06376201
Title: A Clinical Study on the Efficacy and Safety of Amphotericin B Cholesteryl Sulfate Complex for Injection in the Empirical First-line Treatment of Patients With Invasive Fungal Diseases
Brief Title: A Clinical Study on the Efficacy and Safety of ABCD in the Treatment of Patients With Invasive Fungal Disease
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2024-018
Record Dates: First submitted 2024-04-01; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Invasive Fungal Disease
MeSH Terms: conditions — Invasive Fungal Infections | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amphotericin B cholesterol-sulfate complex (ABCD) (Experimental): Investigational drug: Amphotericin B cholesterol-sulfate complex (ABCD) at the same time as a treatment for underlying disease.
  Dosage: According to the patient's condition and the investigator's judgment, the initial dose of ABCD can be 0.5-1.0mg/kg/d, and the dose can be increased daily according to the situation, and the therapeutic dose can be increased to 3.0-4.0mg/kg/d on the third day.
  Course of treatment: ≥ 14 days (whether to continue to receive trial drug treatment after 14 days is decided by the investigator according to the patient's condition).
  Interventions: Drug: Amphotericin B cholesterol-sulfate complex for injection

INTERVENTIONS:
Drug: Amphotericin B cholesterol-sulfate complex for injection — Patients were eligible for enrollment on antifungal therapy with injectable amphotericin B cholesterol-sulfate complex (ABCD) at the same time as a treatment for underlying disease.
  Dosage: According to the patient's condition and the investigator's judgment, the initial dose of ABCD can be 0.5-1.0mg/kg/d, and the dose can be increased daily according to the situation, and the therapeutic dose can be increased to 3.0-4.0mg/kg/d on the third day.
  Course of treatment: ≥ 14 days (whether to continue to receive trial drug treatment after 14 days is decided by the investigator according to the patient's condition).

SUMMARY:
This study is a prospective, multicenter, single-arm study, that aims to evaluate the efficacy and safety of amphotericin B cholesterol-sulfate complex (ABCD) for injection in the first-line treatment of patients with invasive fungal diseases, hoping to provide a reference for the clinical treatment of invasive fungal diseases. Patients with hematologic diseases who meet the criteria for inclusion and discharge with febrile neutropenia and suspected fungal infection were treated with ABCD antifungal therapy for 14 days while receiving treatment for underlying diseases, and the response rate of treatment was observed.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥ 18 years old, gender is not limited;
2. Patients with hematologic malignancies such as leukemia and lymphoma who have undergone chemotherapy or hematopoietic stem cell transplantation;
3. Peripheral blood absolute neutrophil count (ANC) < 0.5×109/L, or expected ANC < 0.5×109/L after 48 h;
4. Within 48 hours before the screening, at least 2 oral temperature measurements (with an interval of more than 30 minutes) ≥ 38.3°C (axillary temperature≥38.0°C), or ≥ 38°C (axillary temperature≥37.7°C) for more than 1h;
5. Received broad-spectrum antimicrobial therapy for at least 96 hours before screening but still had recurrent or persistent fever and suspected fungal infection;
6. The patient or his/her legal representative signs the informed consent form.

Exclusion Criteria:

1. Those who are allergic to amphotericin class B drugs or any component of the cholesterol-sulfate complex;
2. Patients with clinical suspicion of invasive fungal disease who have received antifungal therapy;
3. Patients with clinically diagnosed or confirmed invasive fungal disease (IFD) during the screening period;
4. Patients with abnormal liver function, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 5 times the upper limit of normal (ULN), or ALT or AST > 3 times ULN and total bilirubin > 1.5 times ULN;
5. Patients with reduced renal function, who need or are currently undergoing hemodialysis or peritoneal dialysis;
6. Clinically significant hypokalemia (defined as serum potassium < 3.2 mmol/L, or blood potassium lower than the lower limit of normal while receiving digitalis therapy), and hypokalemia cannot be corrected before starting trial treatment;
7. Expected survival time< 3 months;
8. Pregnant women, lactating women, or women of childbearing age who have not taken contraceptive measures and are planning to become pregnant;
9. Other investigators believe that it is not appropriate to participate in clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Treatment is effective | 12 months
  A patient is considered successful if they meet the following five criteria:
  Starting antifungal treatment until no new fungal infections occur within 7 days after discontinuation of medication; Patient survival within 7 days after discontinuation of treatment; During the treatment period, the drug was not stopped due to side effects or lack of efficacy; After starting antifungal therapy, patients experience fever reduction during neutropenia (defined as body temperature<38 ℃ for more than 48 hours); Invasive fungal diseases diagnosed or clinically diagnosed (baseline fungal infection refers to fungal infection confirmed within 24-48 hours after initiation of antifungal treatment) achieve complete or partial efficacy at the end of treatment.
  Refer to the "Diagnostic Criteria and Treatment Principles for Invasive Fungal Disease in Patients with Hematological Diseases/Malignant Tumors (Sixth Revised Edition)" for the evaluation criteria for the treatment efficacy.

SECONDARY OUTCOMES:
Incidence of the single index in the five criteria of treatment success | 12 months
  The incidence of a single indicator among the five criteria for treatment success mentioned in "Outcome 1"
Completion rate of ABCD treatment for at least 14 days | 12 months
  Completion rate of ABCD treatment for at least 14 days

IPD SHARING:
Plan to Share IPD: No
A summary report will be written and published after the clinical trial is completed, and the data from the summary report or article will be shared

REFERENCES:
- [Result] Sun Y, Huang H, Chen J, Li J, Ma J, Li J, Liang Y, Wang J, Li Y, Yu K, Hu J, Jin J, Wang C, Wu D, Xiao Y, Huang X. Invasive fungal infection in patients receiving chemotherapy for hematological malignancy: a multicenter, prospective, observational study in China. Tumour Biol. 2015 Feb;36(2):757-67. doi: 10.1007/s13277-014-2649-7. Epub 2014 Oct 8. PMID 25293517
- [Result] Sun Y, Meng F, Han M, Zhang X, Yu L, Huang H, Wu D, Ren H, Wang C, Shen Z, Ji Y, Huang X. Epidemiology, management, and outcome of invasive fungal disease in patients undergoing hematopoietic stem cell transplantation in China: a multicenter prospective observational study. Biol Blood Marrow Transplant. 2015 Jun;21(6):1117-26. doi: 10.1016/j.bbmt.2015.03.018. Epub 2015 Mar 31. PMID 25840339
- [Result] Chinese Association Hematologists; Chinese Invasive Fungal Infection Working Group. [The Chinese guidelines for the diagnosis and treatment of invasive fungal disease in patients with hematological disorders and cancers (the 6th revision)]. Zhonghua Nei Ke Za Zhi. 2020 Oct 1;59(10):754-763. doi: 10.3760/cma.j.cn112138-20200627-00624. Chinese. PMID 32987477
- [Result] White MH, Bowden RA, Sandler ES, Graham ML, Noskin GA, Wingard JR, Goldman M, van Burik JA, McCabe A, Lin JS, Gurwith M, Miller CB. Randomized, double-blind clinical trial of amphotericin B colloidal dispersion vs. amphotericin B in the empirical treatment of fever and neutropenia. Clin Infect Dis. 1998 Aug;27(2):296-302. doi: 10.1086/514672. PMID 9709879
- [Result] Dupont B. Clinical efficacy of amphotericin B colloidal dispersion against infections caused by Candida spp. Chemotherapy. 1999 Jun;45 Suppl 1:27-33. doi: 10.1159/000048467. PMID 10394018
- [Result] Gurwith M. Clinical efficacy of amphotericin B colloidal dispersion against infections caused by Aspergillus spp. Chemotherapy. 1999 Jun;45 Suppl 1:34-8. doi: 10.1159/000048468. PMID 10394019
- [Result] Herbrecht R, Letscher-Bru V, Bowden RA, Kusne S, Anaissie EJ, Graybill JR, Noskin GA, Oppenheim, Andres E, Pietrelli LA. Treatment of 21 cases of invasive mucormycosis with amphotericin B colloidal dispersion. Eur J Clin Microbiol Infect Dis. 2001 Jul;20(7):460-6. doi: 10.1007/s100960100528. PMID 11561801
- [Result] Bowden R, Chandrasekar P, White MH, Li X, Pietrelli L, Gurwith M, van Burik JA, Laverdiere M, Safrin S, Wingard JR. A double-blind, randomized, controlled trial of amphotericin B colloidal dispersion versus amphotericin B for treatment of invasive aspergillosis in immunocompromised patients. Clin Infect Dis. 2002 Aug 15;35(4):359-66. doi: 10.1086/341401. Epub 2002 Jul 25. PMID 12145716
- [Result] Dong lu Zhao,Jun Ma. Guiding principle for the administration of amphotericin B colloidal dispersion for injection[J].Journal of Clinical Hematology, 2022, 35(5):6. DOI : 10.13201 / j.issn.1004-2806.2022.05.001.
- See also: Related Info — https://lcxy.whuhzzs.com/data/article/lcxy/preview/pdf/lcxyxzz-35-5-303.pdf